CLINICAL TRIAL: NCT05280873
Title: Clinical Study of Pirfenidone Combined With Methylprednisolone Versus Methylprednisolone in the Treatment of Checkpoint Inhibitor-related Pneumonitis
Brief Title: Pirfenidone Combined With Methylprednisolone Versus Methylprednisolone in the Treatment of CIP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Chengzhi (Other)
Collaborators: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROC202107
Record Dates: First submitted 2021-10-11; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Pneumonitis; Malignant Tumor
Keywords: Pirfenidone; Methylprednisolone
MeSH Terms: conditions — Pneumonia; Neoplasms | interventions — pirfenidone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: We randomly divided the patients into two groups and received pirfenidone combined with methylprednisolone or methylprednisolone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Grade 3-4 checkpoint inhibitor-related pneumonitis
  Interventions: Drug: Pirfenidone, methylprednisolone
- Control group (Experimental): Grade 3-4 checkpoint inhibitor-related pneumonitis
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Pirfenidone, methylprednisolone — Methylprednisolone 2 mg / kg / d+ pirfenidone (starting from 200mg tid, increasing to 600mg tid within one week and maintaining) . Methylprednisolone was reduced according to the researcher's evaluation of the patient's condition and the specific course of treatment was determined.
  Arms: Experimental group
Drug: Methylprednisolone — Methylprednisolone 2 mg / kg / d . Methylprednisolone was gradually reduced after the improvement of symptoms and imaging. The treatment course was 6-8 weeks
  Arms: Control group

SUMMARY:
Checkpoint inhibitor-related pneumonitis (CIP）is a common fatal immune-related adverse event of PD-1/PD-L1 inhibitors. Some CIP patients have poor effect on hormone therapy, and the remission time of CIP varies greatly. Antifibrotic drugs may be effective in patients with CIP.

DETAILED DESCRIPTION:
Pirfenidone can inhibit the occurrence and development of pulmonary fibrosis, reduce pulmonary exudation by inhibiting VEGF and promote pulmonary recovery. In our study, subjects with checkpoint inhibitor-related pneumonitis receive pirfenidone plus methylprednisolone or methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is 18 to 75 years old.
2. Malignant tumors proved by pathology.
3. The subject has received at least one course of immune checkpoint inhibitor treatment.
4. The subject developed grade 3-4 CIP.
5. Take proper contraceptive measures.
6. Appropriate organ system function.
7. Subjects voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. Previous treatment with pirfenidone.
2. Clinically significant hemoptysis occurred within 3 months before enrollment (hemoptysis greater than 50ml per day); Or significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood + + or above, or macrovasculitis.
3. Arteriovenous thrombosis events occurred within 12 months before enrollment, such as cerebrovascular accident, deep venous thrombosis and pulmonary embolism.
4. Abdominal surgery was performed 4 weeks before enrollment, or there was a history of hollow organ perforation.
5. Use nintedanib, cyclophosphamide or cyclosporin within 56 days before enrollment.
6. Suffering from active pulmonary tuberculosis.
7. Patients with mental illness and poor compliance.
8. Sperm / egg donors within 6 months.
9. Lactating women.
10. Persons allergic to pirfenidone.
11. In the investigator's judgment, there are other factors that may have led to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Degradation time of CIP | Approximately 3 months
  According to CTCAE 4.0 and imaging grade of CIP, the time of reduction by one grade was evaluated.
Proportion of degradation within three months | Approximately 3 months
  The number of enrollments reduced by grade 1 in 3 months divided by the total number of enrollments.

SECONDARY OUTCOMES:
Safety(Adverse Events) | From the day the patient signs informed consent form until 30 days after the last medication
  Safety will be assessed according to common terminology criteria for adverse events version 4.0 (CTCAE 4.0)
Total amount of hormone | From the day the patient signs informed consent to the last medication，assessed up to 24 months
  Total amount of methylprednisolone
MMRC score | From the day the patient received treatment until 30 days after the last medication
  Change of Modified Medical Research Council Dyspnea Scale

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, MA, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No plan.